CLINICAL TRIAL: NCT07124052
Title: Comparison of Pain Perception in a Group of Pediatric Patients Undergoing Maxillary Primary Molar Extraction Using a Novel Anesthetic Device Versus Conventional Infiltration: A Randomized Controlled Trial
Brief Title: Comparison of Pain Perception in A Group of Pediatric Patients Undergoing Maxillary Primary Molar Extraction Using A Novel Anesthetic Device Versus Traditional Infiltration
Acronym: SO5PED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Hesham ElSayed Mohamed ElTanahy (Other)
Responsible Party: Sponsor-Investigator, Aya Hesham ElSayed Mohamed ElTanahy, Master's Candidate in Pediatric Dentistry, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8820255
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pain; Extraction, Tooth
Keywords: Pediatric Dentistry; Pain Perception; SleeperOne 5; Computer-Controlled Anesthesia; Conventional Infiltration
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Infiltration (Experimental): Children in this group will receive local anesthesia using the SleeperOne® 5 electronic anesthesia delivery system (Dental Hi-Tec, France). The anesthetic solution used is 3% mepivacaine (Mepecaine-L®, Alexandria Co. for Pharmaceuticals and Chemical Industries, Egypt), administered via the device which controls flow and pressure to minimize discomfort during extraction of maxillary primary molars.
  Interventions: Device: SleeperOne 5
- Conventional Infiltration Technique (Active Comparator): Children in this group will receive local anesthesia using conventional infiltration via a standard dental syringe with a 30-gauge short needle. The anesthetic used is 3% mepivacaine (Mepecaine-L®, Alexandria Co. for Pharmaceuticals and Chemical Industries, Egypt). Buccal infiltration will be administered prior to extraction of maxillary primary molars.
  Interventions: Procedure: (Conventional Infiltration Anesthesia)

INTERVENTIONS:
Device: SleeperOne 5 — A computerized local anesthetic delivery system (manufactured by Dental Hi-Tec, France) designed to minimize pain perception in children during dental procedures by controlling the pressure and flow rate of anesthetic injection. It will be used to deliver 3% mepivacaine (Mepecaine-L®, Alexandria Co. for Pharmaceuticals, Egypt) during maxillary primary molar extraction in pediatric patients.
  Arms: Conventional Infiltration
Procedure: (Conventional Infiltration Anesthesia) — Local anesthetic solution (3% mepivacaine with no vasoconstrictor), manufactured by Alexandria Co. for Pharmaceuticals, Egypt. It will be administered using a 30-gauge short dental needle and standard dental syringe for conventional infiltration anesthesia during primary maxillary molar extraction in pediatric patients.
  Arms: Conventional Infiltration Technique

SUMMARY:
This study aims to compare the pain felt by children during tooth extraction using two different techniques for giving local anesthesia. One group of children will receive anesthesia using a modern electronic device called SleeperOne® 5, which controls the flow and pressure of the anesthesia to reduce pain. The other group will receive anesthesia using the traditional syringe method, which is more commonly used in dental clinics.

The study will include children between the ages of 3 and 5 years old who need to have an upper baby molar tooth extracted. All children in the study will be healthy (classified as ASA I or II), and their parents must agree to participate.

During the procedure, each child will first receive a topical anesthetic gel to numb the surface. Then, based on random selection, the child will receive local anesthesia using either the SleeperOne® 5 device or the traditional syringe. Pain levels during the injection and during the extraction will be measured using special scales suitable for children. Other factors like how long the anesthesia takes to work and how long it lasts will also be recorded.

This research will help dentists understand whether the SleeperOne® 5 device offers a more comfortable experience for young children compared to the traditional method. The goal is to reduce fear and pain during dental treatments for kids.

DETAILED DESCRIPTION:
This randomized controlled clinical trial is designed to evaluate and compare the pain perception in pediatric patients during maxillary primary molar extraction when local anesthesia is administered using either the SleeperOne® 5 electronic delivery system or the conventional infiltration technique with a standard syringe.

Participants will be healthy children aged 3 to 5 years, classified as ASA I or ASA II, requiring extraction of a maxillary primary molar. After obtaining informed consent from the parent or guardian, eligible participants will be randomly assigned to one of two groups using a sealed-envelope technique.

Both groups will receive topical anesthesia prior to local injection. In the control group, local anesthesia will be administered using a traditional 30-gauge dental needle and syringe. In the intervention group, anesthesia will be delivered using the SleeperOne® 5 device, which offers controlled flow and pressure to minimize discomfort.

Pain during injection and during extraction will be evaluated using both subjective and objective pain assessment tools: the Wong-Baker Faces Pain Rating Scale (WBFPR) and the Sound, Eye, Motor (SEM) scale. Secondary outcomes will include time of anesthetic onset and duration, as well as any post-operative complications such as soft tissue trauma or ulceration.

All procedures will be performed by the same pediatric dentist to ensure consistency, and the clinical environment will follow standard infection control protocols. This study aims to determine whether the use of a computer-assisted anesthesia system provides superior comfort and patient experience compared to conventional methods in young children undergoing dental extractions.

ELIGIBILITY:
* Inclusion criteria:

  * Children aged 3-5 years old
  * Medically fit children classified as ASA physical status I and II
  * Parents acceptance to participate in the study (informed consent)
  * Pediatric patients having teeth that have been diagnostically confirmed as requiring extraction.

Exclusion criteria:

* Uncooperative children.
* Patients with an allergy to local anesthesia.
* Children in need of treatment under general anesthesia.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Pain perception during local anesthetic injection | during local anesthetic injection (within 1-2 minutes)
  Pain will be assessed during the injection phase using the Wong-Baker Faces Pain Rating Scale (WBFPRS), a validated tool for pediatric pain assessment. Children will be asked to point to the face that best describes their pain level immediately after the injection is completed.

SECONDARY OUTCOMES:
Effectiveness: Onset and recovery time of local anesthesia | During and immediately after the procedure (Reference: Saoji et al., 2019)
  Effectiveness will be evaluated by recording the time from injection to onset of anesthesia and from completion of the procedure to recovery. Timing will be measured in minutes using a stopwatch.
Duration of the procedure (injecting the anesthesia) | During the procedure (Reference: Saoji et al., 2019)
  The total length of the procedure will be recorded from the start of the anesthetic injection to the completion of tooth extraction. Time will be measured in minutes using a stopwatch.
Incidence of postoperative ulcers | 24 hrs follow up
  The presence or absence of ulcers following the procedure will be evaluated through clinical examination and parental reporting. The outcome will be recorded as a binary value (yes/no).
Pain experienced during extraction | During tooth extraction (Reference: Dhake et al., 2022)
  Pain perception during extraction will be assessed using the Sound, Eye, Motor (SEM) behavior scale. A numerical value will be recorded based on the patient's observed response.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: it introduces the sleeper one 5 anesthetic device — https://www.dentalhitec.com/
- Available data/document: Informed Consent Form: SleeperOne2025 — https://clinicaltrials.gov/study-protocol-pending — Study protocol will be uploaded and publicly accessible upon final approval.